CLINICAL TRIAL: NCT01680510
Title: The Effect of Oral Administration of 9-cis β Carotene Rich Powder of the Alga Dunaliella Bardawil on Visual Functions in Patients With Retinitis Pigmentosa
Brief Title: The Effect of Oral Administration of 9-cis β Carotene Rich Powder of the Alga Dunaliella Bardawil
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Director of Hereditary Retinal Diseases and Electrophysiology Clinic, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-12-9373-YR-CTIL
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Alga vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alga Dunaliella Bardawil 9-cis beta Carotene Rich Powder (Experimental): 50 patients will receive first the capsules containing the alga Dunaliella Bardawil 9-cis beta-Carotene rich powder and after 24 weeks of washout period will receive capsule containing placebo (Starch).
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil; Other: Placebo (starch)
- Placebo (Starch) (Placebo Comparator): The other 50 Patients will receive first the placebo (Starch) capsules and after 24 weeks of washout period will receive capsules containing the alga Dunaliella Bardawil 9-cis beta-Carotene rich powder .
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil; Other: Placebo (starch)

INTERVENTIONS:
Dietary Supplement: Alga Dunaliella Bardawil
Other: Placebo (starch)

SUMMARY:
Retinitis pigmentosa is a genetically disease consisting of progressive retinal degeneration starting in the rods. Its prevalence is 1:4000 people and is the fourth most common blinding disease in Israel in 2004 [7% of all blindness]. The investigators treated a non-progressive form of the disease [Fundus Albipunctatus] by oral therapy of the food supplement made from alga Dunaliella Bardawil composed of approximately 50% 9-cis β-carotene. The alga Dunaliella Bardawil accumulates high concentration of β -carotene when grown under appropriate conditions. The β -carotene of the alga is composed of approximately 50% of all-trans - β carotene and 50% 9-cis β -carotene.

The 9-cis β -carotene has been shown to be a precursor of 9-cis retinoic acid both in-vitro in human intestinal mucosa and in-vivo in a ferret, perfused with 9-cis b-carotene. The night vision, as measured objectively by electroretinography (ERG) more than doubled in six patients tested following treatment. The visual field was also improved significantly. In a more recent study the investigators treated 29 retinitis pigmentosa patients with the 9-cis b Carotene algae Dunaliella Bardawil in a double masked placebo control cross over trial. Significant improvement in retinal function was recorded in 34% of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Men or women aged 18 years or older.
* Electroretinogram (ERG) responses compatible with the diagnosis of Retinitis Pigmentosa

Exclusion Criteria:

* Current smokers.
* Current use of Vitamin A/ beta carotene supplements.
* Active arterial disease within 3 months of study entry such as unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke, and coronary artery bypass graft (CABG) surgery.
* History of malignancy, except basal or squamous cell skin carcinoma.
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception.
* Uncontrolled hypertension defined as either resting diastolic blood pressure of >95mmHg (taken from the mean of 3 readings) or resting systolic blood Pressure of > 180 mmHg.
* History of alcohol abuse or drug abuse, or both.
* Patient plans to engage in vigorous exercise or an aggressive diet regimen.
* Uncontrolled endocrine or metabolic disease.
* Participation in another investigational drug study within 4 weeks of entry into this study.
* Serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Subject whose hormone replacement therapy (HRT) or oral contraceptive therapy (OCT) was initiated within the 3 month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean binocular maximal scotopic electroretinogram b-wave response | At weeks 0, 24,48,72
  Using the protocol of the International Society for Clinical Electrophysiology of Vision and the UTAS 3000 system (LKC Technologies, Gaithersburg, MD), full-field electroretinographic responses will be recorded from both eyes of each patient. For scotopic conditions, maximal ERG b-wave responses will be recorded following 30 minutes of dark adaptation.

SECONDARY OUTCOMES:
The area within the Dark adapted chromatic Goldamann Visual field in isopters in cm2 | at weeks 0, 24, 48, 72
  Kinetic visual field for chromatic stimuli will be recorded in both eyes after 30 minutes of dark adaptation. Area of vision within the isopter will be measured by software in cm2.
The area within Goldamann Visual field in isopters in cm2 | at weeks 0, 24, 48, 72
  Kinetic visual field will be recorded in both eyes. Area of vision within the isopter will be measured by software in cm2.
Mean binocular maximal photopic electroretinogram b-wave response | Weeks 0, 24, 48, 72
  Using the protocol of the International Society for Clinical Electrophysiology of Vision and the UTAS 3000 system (LKC Technologies, Gaithersburg, MD), full-field photopic electroretinographic responses will be recorded from both eyes of each patient.
Best-corrected visual acuity (EDTRS) | Weeks 0, 24, 48, 72

OTHER OUTCOMES:
Objective visual field by chromatic multifocal pupillometer | Weeks 0, 24,48,72
  Objective evaluation of 76 point visual field using a chromatic multifocal pupillometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ygal Rotenstreich, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Rotenstreich Y, Belkin M, Sadetzki S, Chetrit A, Ferman-Attar G, Sher I, Harari A, Shaish A, Harats D. Treatment with 9-cis beta-carotene-rich powder in patients with retinitis pigmentosa: a randomized crossover trial. JAMA Ophthalmol. 2013 Aug;131(8):985-92. doi: 10.1001/jamaophthalmol.2013.147. PMID 23700011
- [Background] Rotenstreich Y, Harats D, Shaish A, Pras E, Belkin M. Treatment of a retinal dystrophy, fundus albipunctatus, with oral 9-cis-beta-carotene. Br J Ophthalmol. 2010 May;94(5):616-21. doi: 10.1136/bjo.2009.167049. Epub 2009 Dec 2. PMID 19955196
- [Background] Skaat A, Sher I, Kolker A, Elyasiv S, Rosenfeld E, Mhajna M, Melamed S, Belkin M, Rotenstreich Y. Pupillometer-based objective chromatic perimetry in normal eyes and patients with retinal photoreceptor dystrophies. Invest Ophthalmol Vis Sci. 2013 Apr 17;54(4):2761-70. doi: 10.1167/iovs.12-11127. PMID 23482470
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764